CLINICAL TRIAL: NCT05977634
Title: The Efficacy of Transcutaneous Tibial Nerve Stimulation on Symptoms of Overactive Bladder and Quality of Life in Women With Idiopathic Overactive Bladder
Brief Title: Transcutaneous Tibial Nerve Stimulation for Idiopathic Overactive Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ege 19-12.3/5
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Overactive Detrusor
Keywords: tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor and investigator that assesses the patients will be blind to the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous tibial nerve stimulation plus bladder training (Experimental): Patients will receive transcutaneous tibial nerve stimulation for 30 minutes, twice a week, for 6 weeks. Application will be done in an outpatient setting, using disposable surface electrodes.
  Interventions: Behavioral: Bladder training; Device: Transcutaneous tibial nerve stimulation
- Bladder training (Other): patients will receive only the routine education program that is given to every patient with idiopathic overactive bladder syndrome. This includes education about the anatomy of the urinary system, patient motivation, and frequent bathroom visits in order to avoid incontinence with gradual increase between each visit to the bathroom.
  Interventions: Behavioral: Bladder training

INTERVENTIONS:
Behavioral: Bladder training — Bladder training has 4 components, educating the patient about anatomy, fluid intake control, pelvic floor muscle contractions and increasing the interval between visits to the bathroom
Device: Transcutaneous tibial nerve stimulation — A combined electrotherapy device capable of applying transcutaneous electrical nerve stimulation will be used. Each session will take 30 minutes. Patient will visit the hospital twice a week for 6 weeks. An electrical current of 0-50 amperes with a frequency of 20 herz, and a duration of 200 micro seconds will be applied using 50x50 mm surface electordes. The aim is to create a tingling sensation without causing any pain on the tibial nerve, at the ankle level.
  Arms: Transcutaneous tibial nerve stimulation plus bladder training

SUMMARY:
This study was designed to assess the efficacy of trans cutaneous tibial nerve stimulation on symptoms of overactive bladder in women with idiopathic overactive bladder

DETAILED DESCRIPTION:
Idiopathic overactive bladder is defined the presence of a sense of urgency with or without accompanying urinary incontinence without an organic pathology or urinary infection. Its prevalence was reported to be between 7.7 to 31 % in women. In this prospective randomized controlled study, we aim to assess the efficacy of trans cutaneous tibial nerve stimulation on symptoms of overactive bladder in women with idiopathic overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Overactive Bladder Questionnaire Validation Study questionnaire 8 scores higher than 11.
* Post voiding residue levels less than 100 ml.
* Women aged between 18-70

Exclusion Criteria:

* Prior history of pelvic surgery
* Pelvic organ prolapsus of grade 2 or more.
* Current urinary tract infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological females will be enrolled in the study.
Enrollment: 26 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Urination frequency | 1 day
  The frequency of urination will be recorded by using a bladder diary. Urination frequency will be questioned before and after the study period.
Severity of overactive bladder symptoms. Overactive Bladder Questionnaire Validation Study questionnaire | 1 day
  This questionnaire assesses the severity of overactive bladder symptoms in 8 items. Each item is scored from 0 to 5. Higher scores denote worse symptom severity. Maximum score is 40. A score over 11 denotes presence of overactive bladder symptoms. Questionnaire will be answered before and after the treatment period.

SECONDARY OUTCOMES:
Quality of life. King's quality of life questionnaire | 1 day
  This questionnaire includes a total of 19 questions assessing general quality of life and also questions related to urinary symptoms. Maximum score is 100 and higher scores denote lower levels of quality of life. Questionnaire will be answered before and after the treatment period.
Level of satisfaction with the treatment. Visual analog scale | 1 day
  After the completion of the study period, patients will be asked to assess their levels of satisfaction with the treatment they received on a visual analog scale.
Incontinence impact questionnaire-7. | 1 day
  This 7 item questionnaire assesses the impact of urinary incontinence on the patients' daily lives. Maximum score is 100. Higher scores denote worse outcomes. Questionnaire will be answered before and after the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Cinar, MD, Principal Investigator — Ege University School of Medicine
Locations (1):
- Ege University School of Medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
May be shared when requested

REFERENCES:
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Int Urogynecol J. 2017 Feb;28(2):191-213. doi: 10.1007/s00192-016-3123-4. Epub 2016 Dec 5. PMID 27921161
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739